CLINICAL TRIAL: NCT06365515
Title: Dopamine and Reward Learning Across Hormonal Transition Phases
Brief Title: Dopamine, Reward Learning and Sex Hormones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Research Foundation (Other); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: TUE010_IRTG_P5
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-08

CONDITIONS: Hormonal Changes; Menstrual Cycle
Keywords: dopamine; fMRI; energy homeostasis; mood homeostasis; sex hormones; motivation; menstrual cycle
MeSH Terms: interventions — benserazide, levodopa drug combination; Levodopa

STUDY DESIGN:
Intervention Model Description: The investigators will assess the effects of Levodopa administration on reward-learning using a double-blind randomized cross-over design. In a within-subject design, participants will get both conditions (Levodopa/placebo) at different time points (a few days apart). After drug/placebo administration we will assess cerebral blood flow and functional connectivity at rest (via functional MR imaging) during effort-based decision making task.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither participants nor investigators will know at which time point the participant will receive Levodopa and placebo tablets. The tablets will be prepared by independent members of the university hospital.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Women in EF (Experimental): Healthy women in the early follicular menstrual cycle phase
  Interventions: Drug: Levodopa administration; Drug: Placebo administration
- Women in ML (Experimental): Healthy women in the mid-luteal menstrual cycle phase
  Interventions: Drug: Levodopa administration; Drug: Placebo administration
- Men (Experimental): Healthy men
  Interventions: Drug: Levodopa administration; Drug: Placebo administration

INTERVENTIONS:
Drug: Levodopa administration — To boost dopamine levels 150mg/37.5 mg L-DOPA/benserazide will be administered in line with recent studies (Kroemer et al., 2019). Maximum plasma concentration of Madopar occur ~60 minutes after drug administration. Participants will start the Effort Allocation Task 45 minutes after Levodopa administration.
  Other Names: Madopar® tablets (Levodopa and Berazidhydrochlorid; Roche)
Drug: Placebo administration — Placebo tablets will be administered as the placebo-controlled condition.
  Other Names: Placebo tablets (P-Tabletten White, Lichtenstein)

SUMMARY:
Hormonal transition periods during the menstrual cycle may predispose women to mental disorders. Hormonal fluctuations provide specific neuroendocrine conditions that modulate brain structure and function and these actions affect cognitive and emotional behaviors and affect energy and mood homeostasis. It is thought that these changes are driven by altered dopamine transmission. Here, the investigators aim to examine (1) how sex hormones and dopamine are linked and also (2) how hormonal changes affect motivation, mood, and energy homeostasis.

To this end, dopamine intervention will be tested on effort-based decision-making and motivational circuits in three hormonal stages (i.e., women in early-follicular phase (EF), women in mid-luteal phase (ML), and men). Additionally, the effects of hormonal status on metabolic indices will be tested, and its effects on mood fluctuations in a period of a month.

The investigator hypothesizes that women in EF cycle phase (1) have naturally less dopamine and show less effort, and (2) they show greater improvement in effort-based decision-making after Levodopa administration. The investigator has exploratory outcomes about (3) sex differences in reward-learning with and without Levodopa administration and explores if these differences correlate with elevated female sex hormone levels. Moreover, it is hypothesized that (4) hormonal fluctuations affect energy homeostasis, thus women in their EF cycle phase have higher energy expenditure and (5) they report more negative mood than in their mid-luteal (ML) cycle phase.

DETAILED DESCRIPTION:
This study will investigate naturally cycling women (n = 60) and men (n = 30). During the intake session (C1) energy expenditure of men and women in their EF cycle phase will be assessed by indirect calorimetry, participants will perform a training EAT task, and hormones (e.g., estradiol, progesterone, testosterone, and their precursor steroids and metabolites) will be assessed from blood samples. Energy expenditure will be assessed at another time point again (C2) (women with different hormonal profiles) and blood samples will be collected.

During the neuroimaging sessions (S1, S2) both men and women will be measured, 30 women in their EF menstrual cycle phase and another 30 women in their ML phase. All participants will take part in the Effort Allocation Task, an effort-based decision-making task during an L-DOPA-based pharmaco-neuroimaging using functional magnetic resonance imaging (fMRI). To disentangle the influence of L-DOPA within a randomized double-blind design, in one session an L-DOPA-based pill (Madopar, 150mg/37.5 mg L-DOPA/ benserazide) and in another one a placebo pill will be administered. Sex steroids (e.g., progesterone, estrogen, testosterone) and metabolic hormones (e.g., glucose, insulin, triglyceride, ghrelin) will be obtained from blood samples. Before and after the MR scanning a reinforcement learning task will be examined.

Over one month, a smartphone survey will be used to regularly record mood, premenstrual symptoms, and information on food cravings. Participants will be asked to start filling out the daily survey after C1 and continue it for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Naturally cycling healthy women and men
* Age between 20-35
* Body-mass index (BMI): 18-28 kg/m2
* German or English language fluency
* Normal or corrected to normal vision
* For women: Regular menstrual cycle, no hormonal contraception (between 25 and 31 days)

Exclusion Criteria:

* Lifetime history of brain injury, stroke, epilepsy, seizures, schizophrenia, bipolar disorders, or severe alcohol/substance dependence, premenstrual dysphoric disorder (anamnestic survey)
* Mood disorder, anxiety disorder, obsessive-compulsive disorder, trauma- and stressor related disorder, somatic symptom disorder or eating disorder in the last 12 months prior to testing (anamnestic survey)
* Severe/uncontrolled medical problems such as hormonal, metabolic, heart or chronic diseases (e.g., severe hypertension, diabetes, dysfunctions of the thyroid, or congestive heart failure)
* Pregnancy, delivery, and lactation (current and within the last year; anamnestic survey)
* Undergoing regular hormonal treatment
* Daily smoking (nicotine, shisha, e-cigarettes) or >1/week (cannabis)
* History of malignant melanoma, angle-closure glaucoma, gastrointestinal ulcers, and osteomalacia
* Hypersensitivity to: Microcrystalline cellulose, Mannitol (Ph.Eur.), Calcium hydrogen phosphate, Pregelatinized Starch (Corn), Crospovidone, Ethylcellulose, Fumed silica, Docusate sodium, Magnesium Stearate (Ph.Eur.), Iron/Ferric oxide (E 172)
* Taking certain types of medication (antihypertensive drugs, sympathomimetics, antipsychotics, drugs affecting the extrapyramidal motor system), non-selective MAO inhibitors or a combination of MAO-A and MAO-B inhibitors
* Since we will only include healthy participants, other medications that might contraindicate Levodopa (e.g., for mental disorders) will be excluded as well. Any other occasional medication will be evaluated on a case-by-case basis.
* Pathological hearing or increased sensitivity to loud noises
* Contraindication for MRI
* Claustrophobia
* Non-removable metal objects on or in the body
* Moderate or severe head injury

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Motivation to work for rewards: force of pressing grip force device (GFD) to gain food and monetary rewards circuitry during effort-based decision-making | During Effort Allocation Task (30 minutes) 45-75 minutes after pharmacological challenge
  Operationalized via the relative force exerted on GFD in an effort allocation task during either the first seconds of each trial (invigoration) or each complete trial (maintenance). Levodopa compared to placebo condition. Outcomes will be compared between groups and will be associated with blood hormone levels.
Reward-related brain responses in the reward network during effort-based decision-making | During task-based neuroimaging (45-75 minutes after drug administration)
  Comparing brain activity (BOLD signals) in response to feedback in regions of the reward network (ROIs: Nucleus Accumbens (NAcc), Putamen, Caudate, Ventral Tegmental Area (VTA), Amygdala, Prefrontal Cortex (PFC), Orbitofrontal cortex (OFC), Anterior Cingulate Cortex (ACC), Insula). Levodopa compared to placebo condition. Outcomes will be compared between groups and will be associated with blood hormone levels.
Reward anticipation on a neural level | During task-based neuroimaging (45-75 minutes after drug administration)
  Comparing brain activity (BOLD signals) in reward-related brain regions (ROIs: NAcc, striatum, PFC, ACC) during the presentation of reward cues with high vs. low reward magnitude after Levodopa administration vs. placebo. Outcomes will be compared between groups and will be associated with blood hormone levels.
Execution of effort on a neural level | During task-based neuroimaging (45-75 minutes after drug administration)
  Comparing brain activity (BOLD signals) in reward-related brain regions (ROIs: Striatum, Insula, ACC, PFC) during force exerted on GFD in an effort allocation task after Levodopa administration vs. placebo. Outcomes will be compared between groups and will be associated with blood hormone levels.

SECONDARY OUTCOMES:
Resting-state functional connectivity | During resting-state neuroimaging (10 minutes)
  Resting-state functional connectivity of regions of the mesocorticolimbic circuitry (ROIs: Nucleus Accumbens, Putamen, Caudata, Ventral Tegmental Area, Amygdala, ventral medial Prefrontal Cortex, Orbitofrontal cortex, Anterior Cingulate Cortex) after Levodopa administration vs. placebo.
Changes in reinforcement learning | During value-based decision-making task (15 minutes) measured 15 minutes before Levodopa administration and 90 min after
  Changes in reward-learning parameters, which are based on choices in the task before Levodopa administration vs. after Levodopa administration and compared to placebo condition.
Menstrual cycle induced changes in mood and food cravings | Measured every day (5 minutes) over the period of one month
  Changes in positive and negative mood ratings (5 mood and 5 stress items, scale 1-10) and in premenstrual symptoms (PSST items, Likert scale 1-4), and in food-craving (FCQ-S items, Likert scale 1-5) measured with ecological momentary assessment.
Changes in resting energy expenditure | Measured twice 1-2 weeks apart, measurement takes 30 minutes
  Menstrual cycle-related changes in resting energy expenditure, measured with indirect calorimetry. Resting energy expenditure will be measured during the early follicular phase and then around ovulation
Changes in metabolic hormone levels during the menstrual cycle | Measured 4 times (5 minutes/day) during a period of 30 days
  Changes in metabolic hormone levels (insulin, glucose, ghrelin, leptin; μg/dL or nmol/L) will be assessed from blood samples during the early follicular phase, ovulatory phase, and mid-luteal phase.

CONTACTS AND LOCATIONS:
Overall Officials: Nils B Kroemer, Professor, Principal Investigator — Department of Psychiatry & Psychotherapy, university of Tübingen
Locations (1):
- Department of Psychiatry & Psychotherapy, University of Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the key results of the study, all anonymized imaging data will be made publicly available (e.g., at openfmri.org)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available after an embargo period of 12 months after completion of the study.
Access Criteria: Until the data is publicly available, researchers may contact the lead PI to gain access.
URL: http://neuromadlab.org